CLINICAL TRIAL: NCT03554122
Title: The Effect of Shotblocker on Pain and Patient Satisfaction for Spinal Anesthesia
Brief Title: Efficacy of Shotblocker in Spinal Needle Related Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Gökhan İNANGİL, Principal Investigator, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SultanAbdulhamid
Record Dates: First submitted 2018-05-26; First posted 2018-06-12 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Needle Phobia; Spinal Anesthesia; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shotblocker Group (Active Comparator): Patients spinal injections were performed with Shotblocker placed onto injection site
  Interventions: Procedure: Shotblocker
- Placebo Group (Placebo Comparator): Patients spinal injections were performed without Shotblocker
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Shotblocker — Patients spinal injections were performed with Shotblocker placed onto injection site
  Arms: Shotblocker Group
Procedure: Placebo — Patients spinal injections were performed without Shotblocker
  Arms: Placebo Group

SUMMARY:
This was a single-blind, randomized controlled trial. Seventy-six patients who underwent spinal anesthesia for surgery were randomized into the Shotblocker group or Control group. Before the insertion of a 25-gauge spinal needle, Shotblocker was applied just before the spinal needle insertion in the Shotblocker group. 10-cm visual analog scale to evaluate the pain intensity of spinal needle insertion and a five-point scale for patient satisfaction were compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery

Exclusion Criteria:

* contraindications to regional anesthesia
* refusal of the patient's regional anesthesia
* intellectual disabilities that prevented completion of a visual analog scale (VAS)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Assessment of pain during spinal needle insertion with 10 cm VAS (Visual Analog Scale) | 2 minutes
  Assessment of pain during spinal needle insertion will be marked on 10 cm VAS scale 0-10 ( 0:no pain 10:Worst possible pain ) by the patient and will be measured

SECONDARY OUTCOMES:
Five point scale for patient satisfaction | 1 minutes
  5 very good, 4 good, 3 satisfactory, 2 unpleasant, 1 very unpleasant
Five point scale for anesthesists satisfaction | 1 minutes
  5 very good, 4 good, 3 satisfactory, 2 unpleasant, 1 very unpleasant

CONTACTS AND LOCATIONS:
Locations (1):
- SBU Sultan Abdulhamid Han, Istanbul, Asia, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Caglar S, Buyukyilmaz F, Cosansu G, Caglayan S. Effectiveness of ShotBlocker for Immunization Pain in Full-Term Neonates: A Randomized Controlled Trial. J Perinat Neonatal Nurs. 2017 Apr/Jun;31(2):166-171. doi: 10.1097/JPN.0000000000000256. PMID 28437308
- [Background] Celik N, Khorshid L. The Use of ShotBlocker for Reducing the Pain and Anxiety Associated With Intramuscular Injection: A Randomized, Placebo Controlled Study. Holist Nurs Pract. 2015 Sep-Oct;29(5):261-71. doi: 10.1097/HNP.0000000000000105. PMID 26263287
- [Background] Cobb JE, Cohen LL. A randomized controlled trial of the ShotBlocker for children's immunization distress. Clin J Pain. 2009 Nov-Dec;25(9):790-6. doi: 10.1097/AJP.0b013e3181af1324. PMID 19851160
- [Background] Drago LA, Singh SB, Douglass-Bright A, Yiadom MY, Baumann BM. Efficacy of ShotBlocker in reducing pediatric pain associated with intramuscular injections. Am J Emerg Med. 2009 Jun;27(5):536-43. doi: 10.1016/j.ajem.2008.04.011. PMID 19497458
- [Background] Koscielniak-Nielsen Z, Hesselbjerg L, Brushoj J, Jensen MB, Pedersen HS. EMLA patch for spinal puncture. A comparison of EMLA patch with lignocaine infiltration and placebo patch. Anaesthesia. 1998 Dec;53(12):1218-22. doi: 10.1046/j.1365-2044.1998.00608.x. PMID 10193230
- [Background] Sharma SK, Gajraj NM, Sidawi JE, Lowe K. EMLA cream effectively reduces the pain of spinal needle insertion. Reg Anesth. 1996 Nov-Dec;21(6):561-4. PMID 8956393